CLINICAL TRIAL: NCT02571634
Title: Open Label Feasibility Pilot Study to Assess the Efficacy and Safety of the Use of Lazanda for Anxiolysis During Radiofrequency Nerve Ablation of Lumbar Facet Joints
Brief Title: Lazanda Fentanyl Nasal Spray Pre Radiofrequency Nerve Ablations(RFA) of Lumbar Facet Joints
Acronym: RFA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Defense and Veterans Center for Integrative Pain Management (Other)
Collaborators: Depomed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 404457
Record Dates: First submitted 2015-10-02; First posted 2015-10-08 (Estimated); Results first posted 2016-10-25 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-07

CONDITIONS: Minor Procedural Pain
Keywords: intranasal fentanyl; conscious sedation
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label (Other): Open label, no blinding, everyone receives Lazanda.
  Interventions: Drug: Lazanda

INTERVENTIONS:
Drug: Lazanda — Given pre radiofrequency ablation of the lumbar facet joints to see if patients can remain alert, and it provides relaxation and pain control.
  Other Names: Intranasal Fentanyl

SUMMARY:
The purpose of this study is to evaluate the effectiveness, feasibility and safety of intranasal fentanyl (Lazanda) as an alternative to the current gold standard (diazepam) to produce anxiolysis and improve patient comfort during and after radiofrequency ablations of the lumbar facet joints. If this pilot study shows a positive effect and Lazanda is found to be feasible and safe for use during procedures, future larger scale studies can be done.

DETAILED DESCRIPTION:
The morning of the procedure/procedures the medication will be obtained from the omnicel by one of the qualified pain clinic study staff for the volunteers that have consented for that day. . It will be signed out on the designated form created for tracking and accountability purposes Patient consent for study participation will be confirmed.

Once in the procedure room a DVPRS (Defense and Veterans Pain Rating Scale) baseline pain score and POSS (Pasero Opioid-induced Sedation Scale) score will be assessed by a member of the research team. Baseline non-invasive blood pressure, heart rate, and oxygen saturation will be documented and continuous monitoring of these vital signs will commence by a provider credentialed by WAMC (Womack Army Medical Center) to perform anxiolysis with documentation every 15 minutes until discharge. A qualified RN (Registered Nurse), or physician will administer 100 mcg of Lazanda ten-fifteen minutes prior to the procedure The administration will be witnessed and confirmed on Appendix D. The unused 7 mcg will be wasted in a charcoal filled bag provided by the manufacturer and that bag will be disposed of per hospital policy. The waste will also be witnessed and noted. The Pasero Opioid-Induced Sedation Scale and a DVPRS pain score will be assessed every 15 minutes through the conclusion of the procedure and every 15 minutes up until discharge or for 1 hour post procedure whichever comes first. If naloxone is required during the procedure this will be noted as well. Any adverse or serious adverse events will be reported per regulatory regulations.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ASA(American Society of Anesthesiologist physical classification system) I-III
* 18 years of age and older Referred for lumbar facet RFA (radio-frequency ablation) by Womack IPMC (Interdisciplinary Pain Management Center)

Exclusion Criteria:

* Known allergy to Fentanyl or naloxone
* Diagnoses of allergic rhinitis with active rhinorrhea
* Pregnant or Breastfeeding
* Asthma or COPD (chronic obstructive pulmonary disease) that requires frequent rescue medications.
* Hepatic insufficiency with abnormal liver enzymes
* Noted decreased mental function
* Heart rate under 50 or BP below 90 systolic and/or 60 diastolic
* Myasthenia gravis diagnoses
* Acute narrow angle glaucoma
* Allergy to meperidine
* On medications with a known dangerous drug interactions to Fentanyl

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael W. Bartoszek, MD, Principal Investigator — Womack Army Medical Center IPMC
Locations (1):
- Womack Army Medical Center, Fort Bragg, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 23 subjects were enrolled between July 20, 2015 and Dec 22, 2015. They were recruited from Womack Army Medical Center's Interdisciplinary Pain Management Center. All were scheduled for a radiofrequency ablation of the lumbar facet joints. All were consented prior to any assessment or treatment.
Period: Overall Study
Arm/Group | Open Label
Started | 23 (First subject wasn't enrolled until July related to receipt of medications from sponsor.)
Completed | 23 (The final subject was enrolled on this date.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Open Label
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 19
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability as Measured by the Number of Adverse Events
Description: Adverse events will be recorded by a yes or no as to their occurence
Time Frame: 24 hours
Measure: Number; unit: adverse events
Groups:
- Open Label: Open label, no blinding, everyone receives Lazanda.
  Lazanda: Given pre radiofrequency ablation of the lumbar facet joints to see if patients can remain alert, and it provides relaxation and pain control.
  There were no adverse events.
Arm/Group | Open Label
Number analyzed (Participants) | 23
adverse events | 0

2. Secondary Outcome: Pain Score Differences Using the DVPRS (Defense and Veterans Pain Rating Scale) Tool.
Description: DVPRS pain scores will be recorded baseline and at 15 minutes post dosing, 30 minutes, 45 minutes and discharge. The DVPRS is a pain scale utilizing color coding descriptive terms and faces to describe pain levels from 0 meaning no pain and 10 the most excruciating pain ever.
Time Frame: Baseline, 15 min, 30 min, 45 min, and discharge
Measure: Mean (Standard Error); unit: pain score
Arm/Group | Open Label
Number analyzed (Participants) | 23
pain score
  Pre procedure average pain score | 4.70 (.31)
  15 minute average pain score | 3.61 (0.42)
  30 minute average pain score | 2.52 (0.50)
  45 minute average pain score | 2.52 (0.43)
  Discharge pain score | 1.65 (0.35)

3. Secondary Outcome: Patient Satisfaction Using a Likert Satisfaction Survey
Description: At 24 hour after the procedure a call was made asking the volunteer to provide a number on a scale to describe their satisfaction with their pain control and their overall satisfaction. A 5 point likert scale was used 1 = very satisfied, 2 satisfied, 3 neither satisfied nor dis-satisfied, 4 not satisfied and 5 very unsatisfied.
Time Frame: 24 hours
Population: Subjects were asked about pain control satisfaction and overall satisfaction using a 5 point likert scale. 1 = very satisfied, 2= satisfied, 3= neither satisfied nor dis-satisfied, 4= not satisfied and 5 = very unsatisfied
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Open Label
Number analyzed (Participants) | 23
Units on scale
  Pain control satisfaction | 1.57 (.15)
  Overall satisfaction | 1.57 (.15)

4. Secondary Outcome: Adverse Events
Description: Volunteers are monitored closely with vs, and sedation levels and any adverse issues will be recorded.
Time Frame: 24 hours
Population: All 23 subjects were monitored with blood pressure, heart rate, oxygen saturation and sedation scores to determine any adverse events.
Measure: Number; unit: number of adverse events
Arm/Group | Open Label
Number analyzed (Participants) | 23
number of adverse events | 0

5. Secondary Outcome: Sedation Level Assessed by POSS Tool
Description: At baseline, 15 minutes post medication receipt, 30 minutes , 45 minutes and at discharge a Pasero-Opioid Sedation Scale Score was obtained. This scale is to measure alertness and amount of sedation. POSS was the abbreviated term used for this scale. The guidelines for that scale include: S= sleeping easily aroused 1= alert and awake; 2= slightly drowsy easily aroused; 3= frequently drowsy, drifts off to sleep during conversation; 4= somnolent, minimal or no response
Time Frame: Baseline, 15 min, 30 min, 45 min, discharge
Measure: Mean (Standard Error); unit: POSS sedation scores
Arm/Group | Open Label
Number analyzed (Participants) | 23
POSS sedation scores
  Pre procedure Poss score | 1 (0)
  Poss score15minutes | 1.04 (.04)
  POSS 30 minutes | 1.04 (.04)
  POSS post 45 minutes | 1.04 (.04)
  POSS discharge | 1.0 (.00)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the initial subject enrolled July 10, 2015 to 24 hours after the final subject on December 22, 2015.
Arm/Group | Open Label
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

LIMITATIONS AND CAVEATS:
This was a pilot study with a small number enrolled without comparison to any other groups. Future studies indicated with larger numbers and comparison to other forms of sedation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No